CLINICAL TRIAL: NCT06888791
Title: Is Hydro Dissection Treatment More Successful With Ultrasonography or Fluoroscopy in the Management of Adhesive Capsulitis?
Brief Title: US-guided Hydro Dissection vs Fluoroscopy-guided Hydro Dissection for Adhesive Capsulitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Supervisor Investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: US-guided vs fluoro-guided HD
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Shoulder Pain
Keywords: Nerve Block; Fluoroscopy; Pain Management
MeSH Terms: conditions — Shoulder Pain; Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US-guided Hydro Dissection (Active Comparator): US-guided hydro dissection for adhesive capsulitis
  Interventions: Procedure: US-guided Hydro Dissection
- Fluoroscopy-guided Hydro Dissection (Active Comparator): Fluoroscopy-guided hydro dissection for adhesive capsulitis
  Interventions: Procedure: Fluoroscopy-guided Hydro Dissection

INTERVENTIONS:
Procedure: US-guided Hydro Dissection — All procedures are performed under sterile conditions. The patient is seated in a sitting position with the physician behind the patient, the shoulder joint and the surrounding area is cleaned extensively with 10% povidone iodine. The probe is placed in the posterior lateral region of the shoulder, below the level of the scapular spine. The posterior labrum is observed as a triangular hyperechoic structure extending from the glenoid to the humeral head. A 22 G spinal needle is inserted approximately 1 cm medial to the probe along the axis of the spina scapula and 8 mg (2 mL) dexamethasone, 80 mg (4 mL) 2% lidocaine, 14 mL 0.9% saline is slowly injected into the joint in a total of 20 mL into the glenohumeral region. For suprascapular nerve block, 2 ml 0.5% bupivacaine + 2 ml 0.9% saline is administered. Patients are followed up in the recovery unit for 30 minutes after the procedure.
  Arms: US-guided Hydro Dissection
Procedure: Fluoroscopy-guided Hydro Dissection — The patient is placed on the scope table in supine position and the shoulder joint is cleaned with 10% povidone iodine. The acromioclavicular joint and the glenohumeral joint are visualized using C-arm fluoroscopy with anteroposterior view. The acromioclavicular joint is marked as the entry point to the shoulder joint. After the skin and subcutaneous tissue is anesthetized with 1 cc 2% lidocaine with a 27 G needle, a 22 G spinal needle is inserted through the acromioclavicular joint and the needle is directed towards the glenohumeral joint. With 1 ml of contrast medium, the localization of the needle is confirmed. After appropriate spread of contrast agent, 8 mg (2 mL) dexamethasone, 80 mg (4 mL) 2% lidocaine, 14 mL 0.9% saline are administered into the joint in a total of 20 mL. For US-guided suprascapular nerve block, 2 ml 0.5% bupivacaine + 2 ml 0.9% saline is administered. Patients are followed up in the recovery unit for 30 minutes after the procedure.
  Arms: Fluoroscopy-guided Hydro Dissection

SUMMARY:
This study aims to evaluate the differences in joint range of motion, Visual Analog Scale (VAS) scores, and the Shoulder Pain and Disability Index (SPADI) outcomes in patients with adhesive capsulitis (frozen shoulder) who undergo hydrodilatation therapy with either ultrasound (USG) or fluoroscopy guidance, in addition to a suprascapular nerve block.

DETAILED DESCRIPTION:
Adhesive capsulitis is a common condition characterized by painful restriction of both active and passive glenohumeral movement, especially when joint degeneration alone is insufficient to explain the limitation. The condition is more prevalent in women and has a strong correlation with diabetes mellitus and thyroid dysfunction. The prevalence in the general population is approximately 3-5%, but it can reach up to 20% in diabetic patients.

The primary goals of treatment are to alleviate pain, improve mobility, shorten symptom duration, and facilitate a return to normal activities. The suprascapular nerve is a major sensory nerve for the posterior and superior aspects of the shoulder and is an accessible target for blockade. Conditions in which suprascapular nerve block is used include chronic shoulder pain syndromes such as rheumatoid arthritis, glenohumeral osteoarthritis, post-stroke shoulder pain, motor neuron disease-related shoulder pain, and various rotator cuff disorders.

Hydrodilatation therapy works by releasing the contracted joint capsule and reducing fibrosis, while corticosteroids exert strong anti-inflammatory effects throughout the shoulder joint. The high-pressure transmission mechanism used in hydrodilatation enhances the distribution of corticosteroids throughout the glenohumeral joint capsule. The procedure involves injecting fluid into the joint cavity under radiological guidance using either ultrasound or fluoroscopy.

This study aims to determine whether performing hydrodilatation under ultrasound versus fluoroscopy guidance in addition to suprascapular nerve block leads to differences in joint range of motion, VAS scores, and SPADI disability index outcomes in patients diagnosed with adhesive capsulitis. Assessments will be performed before the procedure, on the day of the procedure, and at the 3rd month

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of frozen shoulder disease
* VAS>5

Exclusion Criteria:

* Other shoulder diseases that may cause shoulder pain (Rotator cuff tear, clavicle fracture, etc.)
* Allergy to local anesthetics
* History of shoulder surgery in the last 12 months
* Pregnancy
* Coagulopathy or antiplatelet use
* The patient has a mental illness that prevents decision-making

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | Change from baseline to 1st and 3rd month after treatment
  VAS is a scale that can be used measuring pain. Scores range from 0 (no pain) to 10 (the worst pain)

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | Change from baseline to 1st and 3rd month after treatment
  SPADI is a self-report questionnaire developed to evaluate patients with shoulder problems. The pain subscale has 5-items and the disability subscale has 8-items.The total score ranges from 0 to 100, with higher scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Gevher Rabia Genc Perdecioğlu, Study Chair — Diskapi TRH
Locations (1):
- Diskapi Training and Research Hospital, Ankara, Turkey (Türkiye)